CLINICAL TRIAL: NCT07125742
Title: The Effect of Chewing Gum, Fennel Tea, and Ginger Tea Consumption on Intestinal Motility and Postpartum Comfort in Women After Cesarean Section: A Randomized Controlled Trial
Brief Title: Effects of Chewing Gum, Fennel, and Ginger Tea on Intestinal Motility and Comfort After Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Şeyma Çatalgöl, Principal Investigator, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 479-479-26
Record Dates: First submitted 2025-08-06; First posted 2025-08-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Flatulence; Constipation in Postnatal Women
Keywords: Women; Fennel; Chewing Gum; Ginger; Cesarean
MeSH Terms: conditions — Flatulence | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chewing gum (Experimental): Starting 6 hours after cesarean section (following first oral fluid intake), at the 8th and 10th hours: The chewing gum group was asked to chew sugar-free gum for 15 minutes at each time point.
  Interventions: Other: Chewing gum
- Fennel Tea (Experimental): Starting 6 hours after cesarean section (following first oral fluid intake), at the 8th and 10th hours: fennel tea group received 2 g of fennel steeped in 150 ml boiling water for 10 minutes.
  Interventions: Other: Fennel Tea
- Ginger Tea (Experimental): Starting 6 hours after cesarean section (following first oral fluid intake), at the 8th and 10th hours: The ginger tea group received 2 g of fresh ginger steeped in 150 ml boiling water for 10 minutes.
  Interventions: Other: Ginger Tea
- Control Group (No Intervention): No intervention will be applied.

INTERVENTIONS:
Other: Chewing gum — The chewing gum group was asked to chew sugar-free gum for 15 minutes at each time point.
  Arms: Chewing gum
Other: Fennel Tea — Fennel Tea: The fennel tea group received 2 g of fennel steeped in 150 ml boiling water for 10 minutes.
  Arms: Fennel Tea
Other: Ginger Tea — Ginger Tea: The ginger tea group received 2 g of fresh ginger steeped in 150 ml boiling water for 10 minutes.
  Arms: Ginger Tea

SUMMARY:
This randomized controlled trial aims to evaluate the effects of chewing gum, fennel tea, and ginger tea consumption on intestinal motility and postpartum comfort in women following cesarean section.

The primary research questions to be answered are: Do chewing gum, fennel tea, or ginger tea accelerate the onset of bowel sounds after cesarean section? Do these interventions affect the time to first gas passage, defecation, and feeling of hunger? Are there differences among these interventions in terms of their impact on abdominal distension and postpartum comfort? Researchers will compare the effects of the interventions between three groups: chewing gum, fennel tea, and ginger tea.

Participants:

Women who underwent cesarean section and voluntarily agreed to participate in the study.

A total of 96 participants were randomly assigned into three groups of 32 each.

Interventions and procedures:

Starting 6 hours after cesarean section (following first oral fluid intake), at the 8th and 10th hours:

The chewing gum group was asked to chew sugar-free gum for 15 minutes at each time point.

The fennel tea group received 2 g of fennel steeped in 150 ml boiling water for 10 minutes.

The ginger tea group received 2 g of fresh ginger steeped in 150 ml boiling water for 10 minutes.

Bowel sounds were auscultated before and 60 minutes after each intervention. The time of first gas passage, first defecation, and first feeling of hunger was recorded.

Abdominal distension was assessed using a Visual Analog Scale (VAS) six times in total (before and 60 minutes after each intervention).

Postpartum Comfort Scale was applied to all participants at the 12th hour post-cesarean.

All data were collected by the researchers. Randomization was supported by a healthcare professional not involved in the study.

DETAILED DESCRIPTION:
This study was conducted to evaluate the effects of chewing gum, fennel tea, and ginger tea consumption on intestinal motility and postpartum comfort in women following cesarean section. Between November 2024 and August 2025, a randomized controlled trial was carried out with 128 women who met the inclusion criteria and had undergone cesarean delivery. Participants were randomly assigned to four groups (chewing gum, fennel tea, ginger tea, and control; n = 32 per group). Interventions were administered at the 6th, 8th, and 10th hours post-cesarean. The chewing gum group was instructed to chew sugar-free gum for 15 minutes at each time point. In the herbal tea groups, 2 grams of either fennel or fresh ginger were steeped in 150 ml of boiling water for 10 minutes and consumed accordingly.

Bowel sounds were assessed before and 60 minutes after each intervention. Time to first flatus, first defecation, and first feeling of hunger were recorded. Abdominal distension severity was evaluated using a Visual Analog Scale (VAS) a total of six times-before and after each intervention. At the 12th hour postpartum, the Postpartum Comfort Scale was administered to all participants. Data were collected by the researchers, and randomization was supported by a healthcare professional not involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* The participant mother's voluntary participation in the study and provision of written and verbal informed consent,
* Having undergone general anesthesia,
* Having at least basic reading and writing skills,
* Being between 38-42 gestational weeks,
* According to the mother's statement and medical records, having no history of asthma, liver disease, cancer, epilepsy, or similar conditions,
* No history of allergies,
* Body Mass Index (BMI) between 18.50-24.99 kg/m².

Exclusion Criteria:

* The participant mother's unwillingness to continue cooperating in the study,
* Having received spinal anesthesia,
* Being under 18 years of age,
* Being over 45 years of age,
* Inability to chew gum,
* Experiencing nausea or similar side effects during the consumption of fennel or ginger,
* The mother's refusal to consume fennel or ginger tea or to chew gum during the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 128 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-08-16 (Actual); Study Completion 2025-08-16 (Actual)

PRIMARY OUTCOMES:
Assessment of postoperative abdominal distension severity following cesarean section using the Visual Analog Scale (VAS) | Postoperative 6th, 7th, 8th, 9th, 10th, and 11th hours
  In this study, the primary outcome is the determination of the severity of abdominal distension after cesarean section using the Visual Analog Scale (VAS). VAS is a subjective tool frequently used in epidemiological and clinical research to measure the intensity of various symptoms, particularly pain. Its validity and reliability have been previously established. The scale used in this study is the simplest vertical form, 10 cm in length. In other words, the number 0 represents "no abdominal distension", while the number 10 indicates "the worst level of abdominal distension." Using this scale, participants were asked to assess the severity of their abdominal distension.
Evaluation of the time to return of postoperative intestinal motility | Postoperative 48 hour
  Postoperative intestinal motility: In all groups, the times to first bowel movement, first flatus, first defecation, and first sensation of hunger after cesarean section were evaluated.

SECONDARY OUTCOMES:
Assessment of the Postnatal Comfort Scale | Postoperative 12 hour
  Postnatal Comfort:The Postpartum Comfort Scale (PCS) was developed by Karakaplan and Yıldız (2010) to assess postpartum comfort and consists of 34 items. The PCS is a 5-point Likert-type scale, with responses ranging from "strongly agree" (5 points) to "strongly disagree" (1 point) for each item.
  For positively worded statements, "strongly agree" indicates the highest level of comfort (5 points), whereas for negatively worded statements, it reflects a lower level of comfort (1 point). Accordingly, the total score on the scale can range from 34 to 170, with higher scores indicating greater postpartum comfort.
  The scale comprises three subdimensions: physical, psychospiritual, and sociocultural. The Cronbach's alpha coefficient for the overall PCS is 0.78, indicating acceptable internal consistency (Karakaplan & Yıldız, 2010).In this study, it was also used to evaluate postpartum comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma ÇATALGÖL, Dr, Principal Investigator — Uşak University, Faculty of Health Sciences, Department of Nursing
Locations (1):
- Uşak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No